CLINICAL TRIAL: NCT07020767
Title: Effect of Two Different Incision Techniques on Soft and Hard Tissue Outcomes in Immediate Implant Placement in Class II Extraction Sockets of the Esthetic Zone: A Randomized Controlled Clinical Trial
Brief Title: Effect of Two Incision Techniques on Soft and Hard Tissue Outcomes in Immediate Implant Placement in Class II Extraction Sockets of the Esthetic Zone:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Fayoum University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R702
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Immediate Dental Implant; Tooth Extraction; Class II Extraction Sockets; Esthetic Zone Implantology
Keywords: Vestibular socket therapy; Class II extraction sockets; Immediate implant placement; Esthetic zone implants; Dental implant esthetics
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Model Description (Additional Details):
  Participants were randomly assigned in a 1:1 ratio to one of two parallel groups:
  Vestibular Socket Therapy (VST) Group: Minimally invasive implant placement via vestibular access with bone grafting and collagen membrane.
  Flap Elevation Group: Conventional mucoperiosteal flap technique with the same implant and grafting protocol.
  Each surgical site (maximum of two per patient) was independently randomized. Outcome assessors and statisticians were blinded to group allocation to reduce bias. The trial aimed to evaluate differences in esthetic and tissue stability outcomes over a 12-month period.
Who Masked: Outcomes Assessor
Masking Description: The study employed single masking, where the clinical outcome assessors, radiographic evaluators, and statisticians were blinded to group assignments. The operating surgeon was not blinded due to the nature of the surgical procedures. Allocation concealment was ensured using sequentially numbered, opaque, sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Socket Therapy (VST) Group (Experimental): Participants in this group underwent immediate implant placement using Vestibular Socket Therapy (VST). A minimally invasive vestibular incision was made, followed by atraumatic extraction, implant placement (BioHorizons, 30 Ncm), bone grafting with MegaOss™ allograft, and placement of a T-barrier™ collagen membrane. The membrane was stabilized with tacks, and the site was closed with 7/0 nylon sutures. Healing was supported by customized composite healing abutments, and final zirconia crowns were delivered at 3 months.
  Interventions: Procedure: Vestibular Socket Therapy (VST) Group
- Flap Elevation Group (Active Comparator): Participants in this group received immediate implant placement using a conventional mucoperiosteal flap elevation approach. After intrasulcular and vertical incisions, atraumatic extraction was followed by implant placement (BioHorizons, 30 Ncm), grafting with MegaOss™ allograft, and coverage with a T-barrier™ collagen membrane, stabilized with tacks. The site was closed with 7/0 nylon sutures, and healing was supported with customized composite healing abutments. Final zirconia crowns were placed at 3 months.
  Interventions: Procedure: Flap Elevation Group

INTERVENTIONS:
Procedure: Vestibular Socket Therapy (VST) Group — A minimally invasive vestibular incision technique for atraumatic tooth extraction, followed by immediate implant placement using BioHorizons implants. The socket is augmented with MegaOss™ allograft and covered with T-barrier™ collagen membrane, stabilized with membrane tacks. Soft tissue closure is achieved with 7/0 nylon sutures. Customized composite healing abutments are used, and zirconia crowns are delivered at 3 months.
  Arms: Vestibular Socket Therapy (VST) Group
Procedure: Flap Elevation Group — Traditional mucoperiosteal flap elevation with intrasulcular and vertical incisions, followed by atraumatic extraction and immediate implant placement using BioHorizons implants. The socket is grafted with MegaOss™ allograft, covered with T-barrier™ collagen membrane, and stabilized with tacks. The site is closed with 7/0 nylon sutures. Healing abutments and zirconia crowns are applied following the same timeline as the VST group.
  Arms: Flap Elevation Group

SUMMARY:
This randomized controlled clinical trial investigates the effect of two different surgical approaches-Vestibular Socket Therapy (VST) and Flap Elevation Technique-on soft and hard tissue outcomes during immediate implant placement in Class II extraction sockets of the anterior maxilla (esthetic zone). The study enrolled 26 systemically healthy adult patients contributing a total of 48 surgical sites. Each site was randomly assigned to one of the two treatment groups.

The VST group employed a minimally invasive vestibular incision to allow atraumatic extraction, implant placement, bone grafting, and membrane placement while preserving the labial soft tissue and periosteal blood supply. The Flap Elevation group followed a conventional intrasulcular flap approach. In both groups, implants were placed with 30 Ncm torque and augmented with MegaOss™ allograft and a resorbable collagen membrane (T-barrier™).

Clinical and radiographic evaluations were conducted at baseline, 6 months, and 12 months post-loading. Outcomes measured included Pink Esthetic Score (PES), peri-implant probing depth (PD), mucosal level changes, and crestal bone level changes.

DETAILED DESCRIPTION:
Tooth extraction in the anterior maxilla, particularly in the esthetic zone, often leads to substantial resorption of the alveolar ridge, predominantly affecting the thin buccal bone plate. Studies have shown that up to 50% of horizontal ridge width can be lost within 6 months of extraction, compromising both soft tissue contours and the feasibility of future implant placement (Araújo & Lindhe, 2005; Schropp, Wenzel, Kostopoulos, & Karring, 2003). This resorption has profound esthetic and functional implications, especially in patients with high smile lines or thin periodontal biotypes.

To address these challenges, immediate implant placement was introduced to reduce treatment time, preserve socket dimensions, and optimize soft tissue outcomes (Kan, Rungcharassaeng, Umezu, & Kois, 2003; Lang, Pun, Lau, Li, & Wong, 2012). While immediate implants help maintain the overall ridge profile, they do not fully prevent bone remodeling of the buccal plate, which often results in soft tissue recession and compromised esthetic outcomes (Botticelli, Berglundh, Buser, & Lindhe, 2003; Chen & Buser, 2014).

Flap design during implant surgery has been identified as a critical factor influencing peri-implant bone and soft tissue healing. The traditional flap elevation approach provides good visibility but disrupts the periosteal blood supply, increasing the risk of bone resorption and soft tissue shrinkage (Fickl et al., 2008; Jeong et al., 2007). By contrast, flapless surgery preserves the periosteal blood supply and minimizes soft tissue trauma, leading to superior bone preservation and reduced postoperative discomfort (Becker, Goldstein, Becker, & Sennerby, 2005; Oh, Shotwell, Billy, & Wang, 2006). However, flapless techniques carry limitations such as reduced access and increased risk of malpositioning the implant or causing thermal bone damage without adequate irrigation (Choudhary et al., 2023).

To overcome the limitations of both approaches, Vestibular Socket Therapy (VST) was developed as a minimally invasive technique that allows simultaneous atraumatic extraction, implant placement, and socket augmentation through a small vestibular access incision (A. Elaskary et al., 2023). VST preserves the integrity of the labial soft tissues and periosteal blood supply, improves labial bone support, and enables simultaneous use of bone grafts and membranes to enhance both hard and soft tissue outcomes (Ghallab et al., 2023). Clinical trials comparing VST to conventional incisal extraction or partial extraction therapy (PET) have demonstrated comparable or superior outcomes in terms of Pink Esthetic Score (PES), soft tissue volume preservation, and facial bone thickness (A. Elaskary et al., 2023; Hamed et al., 2023).

Bone grafting materials used in combination with immediate implants have also been extensively studied. While autogenous bone has been considered the gold standard, it is often limited by donor site morbidity. Alternatives such as deproteinized bovine bone mineral (DBBM), demineralized bone matrix (DBM), and collagen plugs have been successfully used to fill peri-implant defects and support labial bone regeneration (Araújo & Lindhe, 2005; Artzi, Tal, & Dayan, 2000; Jensen & Terheyden, 2009). Randomized controlled trials have shown that using a combination of autogenous bone chips with DBBM (e.g., MinerOss X) significantly increases facial bone thickness compared to collagen plug or DBM alone (Hamed et al., 2023).

Moreover, the Pink Esthetic Score (PES) has become a standard metric to assess esthetic outcomes around implants, evaluating parameters such as mesial and distal papilla fill, soft tissue level and contour, alveolar process deficiency, and tissue color and texture (Fürhauser et al., 2005). Studies have consistently shown that minimally invasive approaches, like VST and PET, score highly on PES, reflecting superior esthetic outcomes (Cosyn et al., 2011; Evans & Chen, 2008).

Vestibular socket therapy (VST) has emerged as a promising minimally invasive approach for preserving soft and hard tissue architecture during immediate implant placement, particularly in challenging esthetic zones. However, its clinical performance compared to conventional flap elevation remains underexplored. This study aims to evaluate the effectiveness of VST combined with Allograft and collagen membrane in enhancing esthetic outcomes, soft tissue stability, and bone preservation advancing minimally invasive protocols toward more predictable, patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 50 years.

Presence of one or more non-restorable or remaining roots in the maxillary anterior region (canine to canine).

Class II extraction sockets confirmed by CBCT.

Sufficient apical and palatal bone to ensure proper implant positioning and primary stability.

Good compliance with treatment visits and oral hygiene.

Medically healthy with no systemic diseases affecting wound healing or implant success.

Exclusion Criteria:

* Systemic conditions that contraindicate implant or periodontal surgery (e.g., immunocompromised, uncontrolled systemic disease).

Smokers, diabetics, or pregnant/lactating women.

History of chemotherapy or radiotherapy in the head and/or neck region.

Patients on bisphosphonate therapy.

Presence of acute infection at the intended implant site.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score (PES) | 6 and 12 months after prosthetic crown delivery
  The Pink Esthetic Score (PES) evaluates seven soft tissue parameters around implants: mesial papilla, distal papilla, soft tissue level, contour, alveolar process deficiency, tissue color, and texture. Each parameter is scored from 0 (poor) to 2 (ideal), with a total possible score of 14. Higher scores reflect better esthetic outcomes.

SECONDARY OUTCOMES:
Peri-Implant Probing Depth (PD) | 6 and 12 months after prosthetic crown delivery
  Probing depth measured at mesial and distal aspects of the implant using a UNC-15 periodontal probe. Change in depth over time will indicate peri-implant tissue stability.
Peri-Implant Mucosal Level Changes | 6 and 12 months after prosthetic crown delivery
  Vertical soft tissue height changes assessed at mesial papilla, mid-facial, and distal papilla using 3D superimposed intraoral scans. Positive values indicate soft tissue gain; negative values indicate recession.
Crestal Bone Level Changes | 6 and 12 months after prosthetic crown delivery
  Crestal bone thickness on the labial side of the implant measured using CBCT scans. Measurements taken at baseline, 6 months, and 12 months. Changes are calculated to assess bone preservation or loss.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma E.Sayed Hassanein, Study Director — Assistant Professor Of Oral Medicine, Periodontology, Oral Diagnosis
Locations (1):
- Nermeen Nagi, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided